CLINICAL TRIAL: NCT05779488
Title: Effects of Lepidium Meyenii (Maca) Extract Supplementation on Immune Function, Inflammatory Responses, Oxidative Stress After Strenuous Endurance Exercise
Brief Title: Maca in Healthy Subjects After Strenuous Endurance Exercise
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Taipei Medical University (Other)
Collaborators: Panion & BF Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N202103118; MOST110-2410-H-038-013 (Other Grant/Funding Number: National Science and Technology Council)
Record Dates: First submitted 2023-02-20; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Healthy
MeSH Terms: interventions — MacA protein, E coli

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: A double-blind, matched-pair study design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- maca group (Experimental)
  Interventions: Dietary Supplement: maca
- Placebo group (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: maca — 2.25 g of Maca extract, twice per day for 12 weeks
  Other Names: Panion & BF Biotech Inc.
  Arms: maca group
Dietary Supplement: placebo — 2.25 g of starch, twice per day for 12 weeks
  Arms: Placebo group

SUMMARY:
The aim of this study is to investigate Lepidium meyenii (Maca) extract supplementation on exercise-induced responses of the biochemical, and physiological parameters.

DETAILED DESCRIPTION:
Thirty healthy male participants were divided into Maca group (2.25 g of Maca extract, twice per day for 12 weeks) and placebo group (n = 15). All participants conducted a graded exercise test on treadmill to determine the maximal oxygen consumption (VO2max) before and after supplementation, and the speed equivalent to 70% VO2max was conducted for an exhaustive endurance exercise test by treadmill for 1 hours, followed by 90% VO2max until exhaustion.The time to exhaustion, peak oxygen consumption, maximal heart rate and average heart rate will be recorded during the exercise period. Venous blood samples will be drawn before, immediately after, 2-hour after, 4-hour after, and 24-hour after the exhaustive endurance exercise test. Data was analyzed by Two-way mixed design ANOVA.

ELIGIBILITY:
Inclusion Criteria:

-

The volunteers included have conditions as stated below :

1. male adult whose no history of cardiovascular, liver, kidney and diabetes disease
2. no acute sport injury
3. did not participated in any clinical trials or research in the last 3 months before our experiment
4. no supplements were taken during the experimental period
5. were requested to maintain their regular daily life style and avoid alcohol intake

Exclusion Criteria:

-

The volunteers were excluded if they have the situation stated below:

1. history of cardiovascular, liver, kidney and diabetes disease
2. acute sport injury
3. participated in any clinical trials or experimental research in the last 3 months before our experiment
4. taking supplement during the experimental period
5. did not maintain their regular eating habit or drink alcohol

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The sample size is small due to the limited research funding. Additionally, considering the sports ability between men and women is significantly different, there would be a large standard deviation if we include both males and females. Thus our study includes male subjects only.
Enrollment: 50 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Concentration of leukocyte | before exercise
Concentration of leukocyte | immediately after exercise
Concentration of leukocyte | 2-hour after exercise
Concentration of leukocyte | 4-hour after exercise
Concentration of leukocyte | 24-hour after exercise
Concentration of neutrophil | before exercise
Concentration of neutrophil | immediately after exercise
Concentration of neutrophil | 2-hour after exercise
Concentration of neutrophil | 4-hour after exercise
Concentration of neutrophil | 24-hour after exercise
Concentration of lymphocyte | beore exercise
Concentration of lymphocyte | immediately after exercise
Concentration of lymphocyte | 2-hour after exercise
Concentration of lymphocyte | 4-hour after exercise
Concentration of lymphocyte | 24-hour after exercise
Concentration of GSH | before exercise
Concentration of GSH | immediately after exercise
Concentration of GSH | 2-hour after exercise
Concentration of GSH | 4-hour after exercise
Concentration of GSH | 24-hour after exercise
Concentration of CD4+ | before exercise
Concentration of CD4+ | immediately after exercise
Concentration of CD4+ | 2-hour after exercise
Concentration of CD4+ | 4-hour after exercise
Concentration of CD4+ | 24-hour after exercise
Concentration of CD8+ | before exercise
Concentration of CD8+ | immediately after exercise
Concentration of CD8+ | 2-hour after exercise
Concentration of CD8+ | 4-hour after exercise
Concentration of CD8+ | 24-hour after exercise
Concentration of CD19+ | before exercise
Concentration of CD19+ | immediately after exercise
Concentration of CD19+ | 2-hour after exercise
Concentration of CD19+ | 4-hour after exercise
Concentration of CD19+ | 24-hour after exercise
Concentration of CD56+ | before after exercise
Concentration of CD56+ | immediately after exercise
Concentration of CD56+ | 2-hour after exercise
Concentration of CD56+ | 4-hour after exercise
Concentration of CD56+ | 24-hour after exercise
IConcentration of GSSG | before exercise
Concentration of GSSG | immediately after exercise
Concentration of GSSG | 2-hour after exercise
Concentration of GSSG | 4-hour after exercise
Concentration of GSSG | 24-hour after exercise
Concentration of CK-MB | before exercise
Concentration of CK-MB | 2-hour after exercise
Concentration of CK-MB | 4-hour after exercise
Concentration of CK-MB | 24-hour after exercise
Concentration of CK-MB | immediately after exercise
Concentration of TNF-α | before exercise
Concentration of TNF-α | immediately after exercise
Concentration of TNF-α | 2-hour after exercise
Concentration of TNF-α | 4-hour after exercise
Concentration of TNF-α | 24-hour after exercise
Concentration of IL-1β | before exercise
Concentration of IL-1β | immediately after exercise
Concentration of IL-1β | 2-hour after exercise
Concentration of IL-1β | 4-hour after exercise
Concentration of IL-1β | 24-hour after exercise
Concentration of IFN-γ | before exercise
Concentration of IFN-γ | immediately after exercise
Concentration of IFN-γ | 2-hour after exercise
Concentration of IFN-γ | 4-hour after exercise
Concentration of IFN-γ | 24-hour after exercise
Concentration of IL-2 | before exercise
Concentration of IL-2 | immediately after exercise
Concentration of IL-2 | 2-hour after exercise
Concentration of IL-2 | 4-hour after exercise
Concentration of IL-2 | 24-hour after exercise
Concentration of IL-4 | before exercise
Concentration of IL-4 | immediately after exercise
Concentration of IL-4 | 2-hour after exercise
Concentration of IL-4 | 4-hour after exercise
Concentration of IL-4 | 24-hour after exercise
Concentration of IL-8 | before exercise
Concentration of IL-8 | immediately after exercise
Concentration of IL-8 | 2-hour after exercise
Concentration of IL-8 | 4-hour after exercise
Concentration of IL-8 | 24-hour after exercise
Concentration of IL-10 | before exercise
Concentration of IL-10 | immediately after exercise
Concentration of IL-10 | 2-hour after exercise
Concentration of IL-10 | 4-hour after exercise
Concentration of IL-10 | 24-hour after exercise
Concentration of TBARS | before exercise
Concentration of TBARS | immediately after exercise
Concentration of TBARS | 2-hour after exercise
Concentration of TBARS | 4-hour after exercise
Concentration of TBARS | 24-hour after exercise
Concentration of PC | before exercise
Concentration of PC | immediately after exercise
Concentration of PC | 2-hour after exercise
Concentration of PC | 4-hour after exercise
Concentration of PC | 24-hour after exercise
Concentration of SOD | before exercise
Concentration of SOD | immediately after exercise
Concentration of SOD | 2-hour after exercise
Concentration of SOD | 4-hour after exercise
Concentration of SOD | 24-hour after exercise
Concentration of catalase | before exercise
Concentration of catalase | immediately after exercise
Concentration of catalase | 2-hour after exercise
Concentration of catalase | 4-hour after exercise
Concentration of catalase | 24-hour after exercise
Concentration of GPx | before exercise
Concentration of GPx | immediately after exercise
Concentration of GPx | 2-hour after exercise
Concentration of GPx | 4-hour after exercise
Concentration of GPx | 24-hour after exercise
Concentration of CK | before exercise
Concentration of CK | immediately after exercise
Concentration of CK | 2-hour after exercise
Concentration of CK | 4-hour after exercise
Concentration of CK | 24-hour after exercise
Concentration of LDH | before exercise
Concentration of LDH | immediately after exercise
Concentration of LDH | 2-hour after exercise
Concentration of LDH | 4-hour after exercise
Concentration of LDH | 24-hour after exercise
Concentration of IL-6 | before exercise
Concentration of IL-6 | immediately after exercise
Concentration of IL-6 | 2-hour after exercise
Concentration of IL-6 | 4-hour after exercise
Concentration of IL-6 | 24-hour after exercise
Concentration of cTnI | before exercise
Concentration of cTnI | immediately after exercise
Concentration of cTnI | 2-hour after exercise
Concentration of cTnI | 4-hour after exercise
Concentration of cTnI | 24-hour after exercise
Concentration of NT proBNP | before exercise
Concentration of NT proBNP | immediately after exercise
Concentration of NT proBNP | 2-hour after exercise
Concentration of NT proBNP | 4-hour after exercise
Concentration of NT proBNP | 24-hour after exercise
Concentration of testosterone | before exercise
Concentration of testosterone | immediately after exercise
Concentration of testosterone | 2-hour after exercise
Concentration of testosterone | 4-hour after exercise
Concentration of testosterone | 24-hour after exercise
Concentration of LH | before exercise
Concentration of LH | immediately after exercise
Concentration of LH | 2-hour after exercise
Concentration of LH | 4-hour after exercise
Concentration of LH | 24-hour after exercise
Concentration of FSH | before exercise
Concentration of FSH | immediately after exercise
Concentration of FSH | 2-hour after exercise
Concentration of FSH | 4-hour after exercise
Concentration of FSH | 24-hour after exercise
Concentration of NO | before exercise
Concentration of NO | immediately after exercise
Concentration of NO | 2-hour after exercise
Concentration of NO | 4-hour after exercise
Concentration of NO | 24-hour after exercise
Concentration of GOT | before exercise
Concentration of GOT | immediately after exercise
Concentration of GOT | 2-hour after exercise
Concentration of GOT | 4-hour after exercise
Concentration of GOT | 24-hour after exercise
Concentration of GPT | before exercise
Concentration of GPT | immediately after exercise
Concentration of GPT | 2-hour after exercise
Concentration of GPT | 4-hour after exercise
Concentration of GPT | 24-hour after exercise
Concentration of BUN | before exercise
Concentration of BUN | immediately after exercise
Concentration of BUN | 2-hour after exercise
Concentration of BUN | 4-hour after exercise
Concentration of BUN | 24-hour after exercise
Concentration of creatinine | before exercise
Concentration of creatinine | immediately after exercise
Concentration of creatinine | 2-hour after exercise
Concentration of creatinine | 4-hour after exercise
Concentration of creatinine | 24-hour after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan